CLINICAL TRIAL: NCT03891108
Title: A Randomized, Open Label, Parallel Design, Single Continuous Intravenous Infusion Study of BMS-986231 to Assess the Pharmacokinetics, Safety and Tolerability of Multiple Formulations in Healthy Participants
Brief Title: A Pharmacokinetics, Safety and Tolerability Study of Multiple Formulations of BMS-986231 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CV013-038
Record Dates: First submitted 2019-03-25; First posted 2019-03-26 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Treatment A: BMS-986231 Formulation A (Active Comparator): Participants will be administered Treatment A: BMS-986231 Formulation A as a 48-hour IV infusion on Day 1, followed by review of safety and tolerability data during and after the infusion.
  Interventions: Drug: BMS-986231 Formulation A
- Treatment B: BMS-986231 Formulation B (Experimental): Participants will be administered Treatment B: BMS-986231 Formulation B as a 48-hour IV infusion on Day 1, followed by review of safety and tolerability data during and after the infusion.
  Interventions: Drug: BMS-986231 Formulation B
- Treatment C: BMS-986231 Formulation C (Experimental): Participants will be administered Treatment C: BMS-986231 Formulation C as a 48-hour IV infusion on Day 1, followed by review of safety and tolerability data during and after the infusion.
  Interventions: Drug: BMS-986231 Formulation C
- Treatment D: BMS 986231 Formulation D (Experimental): Participants will be administered Treatment D: BMS 986231 Formulation D as a 48-hour IV infusion on Day 1, followed by review of safety and tolerability data during and after the infusion.
  Interventions: Drug: BMS-986231 Formulation D

INTERVENTIONS:
Drug: BMS-986231 Formulation A — Participants will be administered BMS-986231 Formulation A as IV infusion for 48 hours.
  Arms: Treatment A: BMS-986231 Formulation A
Drug: BMS-986231 Formulation B — Participants will be administered BMS-986231 Formulation B as IV infusion for 48 hours.
  Arms: Treatment B: BMS-986231 Formulation B
Drug: BMS-986231 Formulation C — Participants will be administered BMS-986231 Formulation C as IV infusion for 48 hours.
  Arms: Treatment C: BMS-986231 Formulation C
Drug: BMS-986231 Formulation D — Participants will be administered BMS-986231 Formulation D as IV infusion for 48 hours.
  Arms: Treatment D: BMS 986231 Formulation D

SUMMARY:
Main Objective of this study is to compare the single intravenous (IV) infusion pharmacokinetics (PK) of BMS-986231 and its metabolites (BMT-284730, BMT-279554, and CAR-000463) following of up to 2 test formulations of BMS-986231 relative to the reference formulation.

DETAILED DESCRIPTION:
Participants will be randomized 1:1:1:1 and dosed with either of the 4 treatments: A, B, C, or D; followed by review of safety and tolerability data during and after the infusion. The study will proceed with treatments A, and C unless one or more of these treatments shows poor tolerability; in which case the study may proceed with treatment B or D in the follow-up cohorts. Additional participants will be randomized equally to each of the treatments the study will proceed with.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be willing to participate in the study and sign the informed consent form (ICF).
* Participants must be willing and able to complete all study-specific procedures and visits.
* Healthy participant, as determined by no clinically significant deviation from normal in medical history, physical examination, ECGs, and clinical laboratory determinations in the opinion of the investigator.
* Body mass index of 18.0 to 32.0 kg/m2, inclusive, and body weight ≥ 45 kg and ≤ 110 kg, at screening.
* Heart rate > 45 bpm and < 95 bpm at screening or baseline (within 30 minutes prior to randomization).
* Systolic BP > 110 mmHg and < 140 mmHg at screening or baseline (within 30 minutes prior to randomization).
* Normal renal function at screening as evidenced by an estimated glomerular filtration rate > 80 mL/min/1.732 calculated with the Chronic Kidney Disease Epidemiology Collaboration formula.
* Males and females, ages 18 or local age of majority to 40 years, inclusive.

Exclusion Criteria:

* Any significant acute or chronic medical illness
* Diagnosis of fibromyalgia
* History of syncope, orthostatic instability, or recurrent dizziness
* History or family history of ocular disorders (eg, glaucoma)
* History of bleeding diathesis (unusual susceptibility to bleed [hemorrhage] mostly due to hypocoagulability)
* Personal history or strong family history of sudden cardiac death, myocardial infarction, or other heart disease considered to be clinically significant by the investigator
* Any major surgery within 4 weeks of study drug administration
* History of Gilbert's Syndrome

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2019-02-28 (Actual); Primary Completion 2019-07-29 (Actual); Study Completion 2019-07-29 (Actual)

PRIMARY OUTCOMES:
Maximum Plasma Concentration (Cmax) of BMS-986231 and its Metabolites (BMT-284730, BMT-279554, and CAR-000463) | Day 1 to Day 5
  Cmax is the maximum plasma concentration.
Average Concentration Over a Dosing Interval (Css-av) of BMS-986231 and its Metabolites (BMT-284730, BMT-279554, and CAR-000463) | Day 1 to Day 5
  Css-av is defined as the average concentration over a dosing interval.
Area Under the Plasma Concentration-Time Curve From Time 0 (Dosing) Extrapolated to Infinity (AUC(INF)) of BMS-986231 and its Metabolites (BMT-284730, BMT-279554, and CAR-000463) | Day 1 to Day 5
  AUC(INF) is defined as area under the plasma concentration-time curve from time 0 (dosing) extrapolated to infinity.
Area Under the Concentration-Time Curve From Time 0 (Dosing) to the Time of the Last Quantifiable Concentration Observed (AUC(0-T)) of BMS-986231 and its Metabolites (BMT-284730, BMT-279554, and CAR-000463) | Day 1 to Day 5
  AUC(0-T) is defined as area under the concentration-time curve from time 0 (dosing) to the time of the last quantifiable concentration observed (T).
Terminal Elimination Phase Half-Life (T-HALF) of BMS-986231 and its Metabolites (BMT-284730, BMT-279554, and CAR-000463) | Day 1 to Day 5
  T-HALF is terminal elimination phase half-life.
Time to Reach Cmax in Plasma (Tmax) of BMS-986231 and its Metabolites (BMT-284730, BMT-279554, and CAR-000463) | Day 1 to Day 5
  Tmax is defined as time to reach Cmax in plasma.
Metabolite to Parent Molar Ratio of AUC(INF) (MRAUC[INF]) and Metabolite to Parent Molar Ratio of Css-av (MRCssav) of Metabolites of BMS-986231 (BMT-284730, BMT-279554, and CAR-000463) | Day 1 to Day 5
  MRAUC(INF) is determined using AUC(INF) for metabolite / AUC(INF) for BMS-986231. MRCss-av is determined using Css-av for metabolite / Css-av for BMS-986231.
Total Systemic Clearance (CLT) of BMS-986231 | Day 1 to Day 5
  CLT is total systemic clearance.
Apparent Volume of Distribution During the Terminal Phase (Vz) of BMS-986231 | Day 1 to Day 5
  Vz is apparent volume of distribution during the terminal phase.
Volume of Distribution at Steady State (Vss) of BMS-986231 | Day 1 to Day 5
  Vss is volume of distribution at steady state.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events (AEs) | Day 1 up to Day 13
  An AE is defined as any new untoward medical occurrence or worsening of a preexisting medical condition in a clinical investigation participant administered study drug and that does not necessarily have a causal relationship with this treatment.
Number of Participants with Serious AEs (SAEs) | From signature of informed consent up to 30 days post last treatment
  A SAE is any untoward medical occurrence that at any dose: results in death, is life-threatening, requires inpatient hospitalisation or prolongation of existing hospitalisation, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, or is an important medical event (defined as a medical event(s) that may not be immediately life threatening or result in death or hospitalization but, based upon appropriate medical and scientific judgment, may jeopardize the participant or may require intervention).
Number of Participants With Significant Changes in Clinical Laboratory Values | Day 1 up to Day 13
  Serology (includes hepatitis C antibody, hepatitis B surface antigen, and human immunodeficiency virus [HIV]-1 and -2 antibody), Hematology and Serum Chemistry (includes C-reactive protein and fibrinogen), Follicle-Stimulating Hormone (FSH) on blood samples, and urinalysis will be performed as part of clinical lab tests.
Number of Participants with Significant Changes in Vital Signs | Day 1 up to Day 13
  Vital signs include body temperature, respiratory rate, and semi-supine blood pressure, and heart rate.
Number of Participants with Significant Changes in Electrocardiograms (ECGs) | Day 1 up to Day 13
  A reflex 12-lead ECG will be conducted to confirm any significant changes in ECGs.
Number of Participants with Significant Changes in Physical Examinations | Day 1 up to Day 13
  The full physical examination will include general appearance, head, eyes, ears, nose, throat, neck, lungs, heart, abdomen, extremities, peripheral pulses, skin, and neurologic examination. Targeted physical exams will include general appearance, oral mucosa, heart, lungs, abdomen, and skin.

CONTACTS AND LOCATIONS:
Locations (1):
- PRA Health Sciences, Salt Lake City, Utah, United States

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm